CLINICAL TRIAL: NCT05700903
Title: Autonomic and Renal Contributions to Hypertension With Androgen Deprivation Therapy
Brief Title: Contributions to Hypertension With Androgen Deprivation Therapy
Acronym: ARCH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 22-2201.cc
Record Dates: First submitted 2023-01-10; First posted 2023-01-26 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Androgen Deprivation Therapy; Prostate Cancer; Hypertension; Autonomic Dysfunction; Renal Disease
MeSH Terms: conditions — Prostatic Neoplasms; Hypertension; Primary Dysautonomias; Kidney Diseases | interventions — Leuprolide; Goserelin; Receptors, Androgen; bicalutamide; Flutamide; enzalutamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Prostate Cancer (Active Comparator): Men undergoing androgen deprivation therapy via gonadotropin releasing hormone agonist plus androgen receptor inhibitor for the treatment of prostate cancer
  Interventions: Drug: Gonadotropin Releasing Hormone Agonists (GNRH); Drug: Androgen receptor (AR) inhibitor
- Healthy + ADT (Active Comparator): Healthy men undergoing gonadal suppression via gonadotropin releasing hormone agonist plus androgen receptor inhibitor for 9 weeks
  Interventions: Drug: Gonadotropin Releasing Hormone Agonists (GNRH); Drug: Androgen receptor (AR) inhibitor
- Healthy + Placebo (Placebo Comparator): Healthy men undergoing placebo for 9 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gonadotropin Releasing Hormone Agonists (GNRH) — 8 weeks of GnRH agonist
  Other Names: Leuprolide; Goserelin
  Arms: Healthy + ADT; Prostate Cancer
Drug: Androgen receptor (AR) inhibitor — 2 weeks of AR Inhibitor
  Other Names: Bicalutamide; Flutamide; Enzalutamide
  Arms: Healthy + ADT; Prostate Cancer
Drug: Placebo — Placebo tablet and injection
  Arms: Healthy + Placebo

SUMMARY:
This study plans to learn more about contributors to high blood pressure in men who undergo androgen deprivation therapy (ADT) to treat prostate cancer. Prostate cancer is the most common non-skin cancer in men, affecting approximately 1 in 8 American men and its primary treatment is through the use of ADT. However, ADT increases the likelihood of developing heart disease including high blood pressure. This study will determine if dysfunction of the nervous system and/or kidneys occurs in men undergoing ADT, as these systems play a significant role in control of blood pressure. The results from this study will help us understand the ways in which ADT contributes to heart disease and help us develop therapies to prevent heart disease in prostate cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* -age 40+ years;
* resting blood pressure <140/90 mmHg;
* fasted blood glucose <126 mg/dL;
* testosterone ≥400 ng/dL;
* sedentary to recreationally active;
* nonsmokers;
* healthy as determined by medical history, physical exam, blood and urine chemistries and resting and exercise ECG during a physician supervised graded exercise treadmill test OR recent diagnosis of non-metastatic prostate cancer with plans to undergo androgen deprivation therapy;
* PSA <4.00 ng/dL if in the non-cancer group;
* Gleason Score ≤7 if in the prostate cancer group;
* no use of medications that might influence cardiovascular function (e.g., antihypertensives, lipid-lowering medications);
* willing and able to be on GnRHagonist and AR inhibitor;
* not taking antioxidant vitamins, corticosteroids, or anti-inflammatory medications, or willing to stop use for four weeks prior to the start of the study;
* not using exogenous sex hormones for at least one year

Exclusion Criteria:

* -acute liver disease;
* chronic kidney disease, serum creatinine >1.3 mg/dL, macroalbuminuria >300 mg/g of proteinuria
* pre-existing or active cardiac, renal or hepatic disease, epilepsy or other seizure disorder;
* diabetes, active or chronic infection, disease that affects the nervous system;
* Gleason Score ≥8;
* thyroid dysfunction, defined as ultrasensitive TSH <0.5 or >5.0 mU/L, volunteers with abnormal TSH values will be re-considered for participation after follow-up evaluation by the PCP with initiation or adjustment of thyroid hormone replacement;
* tobacco use within the previous 12 months

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Change in Cardiovagal Baroreflex Sensitivity | Before and after 9 weeks of androgen deprivation therapy or placebo
  The change in cardiovagal baroreflex sensitivity will be assessed the modified Oxford procedure
Change in blood pressure reactivity to the cold pressor test | Before and after 9 weeks of androgen deprivation therapy or placebo
  The change in blood pressure will be assessed from quiet rest to sympathetic activation using the cold pressor test
Change in exercise pressor reflex | Before and after 9 weeks of androgen deprivation therapy or placebo
  The change in blood pressure will be assessed from quiet rest to isometric handgrip exercise
Change in ambulatory blood pressure variability | Before and after 9 weeks of androgen deprivation therapy or placebo
  Ambulatory blood pressure variability will be determined from 24-hour ambulatory blood pressure monitoring.
Change in beat-to-beat blood pressure variability | Before and after 9 weeks of androgen deprivation therapy or placebo
  Beat-to-beat blood pressure variability will be using finger photoplethysmography measured in the laboratory.
Change in renal vascular resistance | Before and after 9 weeks of androgen deprivation therapy or placebo
  Renal blood flow will be determined using ultrasound and blood pressure will be determined using finger photoplethysmography. These measures will be used to estimate renal vascular resistance.
Change in Renal dysfunction biomarkers | Before and after 9 weeks of androgen deprivation therapy or placebo
  Neutrophil gelatinase-associated lipocalin (NGAL), kidney injury molecule (KIM)-1, interleukin (IL)-18, and vanin-1 will be quantified in urine using commercially available assay kits. Concentrations will be normalized to urinary flow rate.

SECONDARY OUTCOMES:
Change in sympathetic baroreflex sensitivity | Before and after 9 weeks of androgen deprivation therapy or placebo
  Changes in muscle sympathetic nerve activity in response to changes in blood pressure will be assessed using the modified Oxford procedure
Change in Sympathetic reactivity | Before and after 9 weeks of androgen deprivation therapy or placebo
  The change in muscle sympathetic nerve activity will be assessed from quiet rest to sympathetic activation using the cold pressor test.
Change in glomerular filtration rate | Before and after 9 weeks of androgen deprivation therapy or placebo
  Glomerular filtration rate and renal plasma flow will be calculated by iohexol (Omnipaque 300, GE Healthcare) clearance technique. Plasma and urine iohexol and p-aminohippurate clearance will be measured on a High-Performance Liquid Chromatography (HPLC, Waters, Milford, MA).
Change in renal plasma flow | Before and after 9 weeks of androgen deprivation therapy or placebo
  Renal plasma flow will be calculated by p-aminohippurate (Basic Pharma) clearance techniques. Plasma and urine p-aminohippurate clearance will be measured on a High-Performance Liquid Chromatography (HPLC, Waters, Milford, MA).

OTHER OUTCOMES:
Change in Inflammation | Before and after 9 weeks of androgen deprivation therapy or placebo
  Proteomic analysis of inflammatory cascade proteins will be quantified in plasma samples.
Change in Oxidative stress | Before and after 9 weeks of androgen deprivation therapy or placebo
  Whole blood reactive oxygen species will be measured in from venous blood samples using electron paramagnetic resonance spectroscopy
Change in Body composition | Before and after 9 weeks of androgen deprivation therapy or placebo
  Descriptive variable total body fat mass (for screening and to document any changes with the intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Babcock, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- UCHealth University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No